CLINICAL TRIAL: NCT02527785
Title: Phase II Study of S-1 in Combination With Oxaliplatin and Irinotecan in Patients With Advanced, Recurrent or Metastatic Gastric Cancer
Brief Title: Study of Oxaliplatin, Irinotecan, and S-1 in Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMC-HO-GI-1401
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Stomach Neoplasm
Keywords: stomach neoplasm; oxaliplatin; irinotecan; S-1
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Irinotecan; S 1 (combination); titanium silicide; Tegafur; gimeracil; Oxonic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin, Irinotecan, S-1(OIS) (Experimental): triple combination with oxaliplatin, irinotecan, and S-1.
  Treatment will be delivered as a 2-week cycle.
  1. Oxaliplatin 65 mg/m2 iv on day 1
  2. Irinotecan 135 mg/m2 iv on day 1
  3. S-1 80 mg/m2/day on day 1-7
  Interventions: Drug: Oxaliplatin, Irinotecan, S-1(OIS)

INTERVENTIONS:
Drug: Oxaliplatin, Irinotecan, S-1(OIS) — Treatment will be delivered every 2 weeks
  1. oxaliplatin 65 mg/m2 iv on day 1
  2. irinotecan 135 mg/m2 iv on day 1
  3. S-1 80 mg/m2/day po on day 1-7
  Other Names: Liplatin, Inotecan, TS-1 (tegafur, gimeracil, oteracil)

SUMMARY:
This study will conduct a phase II study of triple combination with oxaliplatin, irinotecan, and S-1 as the first-line chemotherapy in patients with advanced gastric cancer.

DETAILED DESCRIPTION:
It is widely accepted that the efficacy of chemotherapy for patients with inoperable, advanced, and metastatic gastric cancer is better than that compared to best supportive care. In general, combination chemotherapies are more efficient than monotherapy and so it is reasonable to give combination chemotherapy to patients with good performance status.

Especially dual combination chemotherapy with fluoropyrimidine and platinum has shown the objective response rate of 25-48% in patients with newly diagnosed advanced metastatic gastric cancer and several studies about triple combination with oxaliplatin, irinotecan, and fluoropyrimidine have shown the response rate of 53~75% but also higher rate of hematologic adverse events. So the investigators had conducted the phase I study of these three drugs with modification of dosage and schedule and will conduct a phase II study with recommended dose of triple chemotherapy from this phase I study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed advanced, recurrent or metastatic adenocarcinoma of stomach (stage IV by primary tumor, regional nodes, metastasis(TNM) staging system)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* More than 3 months expected life span
* Measurable lesion by RECIST criteria version 1.1
* Palliative chemotherapy naive
* Adequate organ functions
* Participants must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* Positive Her2 status on participants' cancer tissue.
* Any prior 2 years or concurrent malignancy other than non-melanoma skin cancer, in situ cancer of uterine cervix, or papillary or follicular thyroid cancer.
* Participants who had received radiation therapy for target lesions 4 weeks before study enrollment
* Participants who had received major surgery 4 weeks before study enrollment
* Participants with active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus, myocardial infarction during the preceding 12 months, pregnancy, or breast feeding
* Participants with central nervous system(CNS) metastases
* Participants with peripheral sensory neuropathies with impaired functional activities
* Participants with gastrointestinal obstruction or bleeding inducing mal-absorption of oral chemotherapeutic agents.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
overall response rate | 1.5 years
  Tumor response will be classified on the basis of the response evaluation criteria in solid tumors (RECIST) guidelines version 1.1

SECONDARY OUTCOMES:
progression free survival | 1.5 years
  The progression-free survival (PFS) will be measured from the start of study treatment until documented tumor progression (by RECIST) or death due to any cause
overall survival | 1.5 years
  The overall survival (OS) will be estimated from the start of study treatment until participant's death and measured using the Kaplan-Meier method
Toxicity profiles - The number of participants and grade of intensity of treatment related adverse events | 1.5 years
  adverse events will be graded using the NCI common terminology criteria for adverse events (NCTCAE) v 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym university medical center, Anyang, Gyunggi, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim HS, Ryu MH, Zang DY, Park SR, Han B, Kang WK, Rha SY, Jung M, Kim JS, Kang BW, Lee KH, Rho SY, Kim JH, Kim KC, Cho JW, Choi DR, Lim H, Kang HS, Soh JS, Kim MJ, Seo J, Kang YK. Phase II study of oxaliplatin, irinotecan and S-1 therapy in patients with advanced gastric cancer: the Korean Cancer Study Group ST14-11. Gastric Cancer. 2018 Sep;21(5):802-810. doi: 10.1007/s10120-018-0794-1. Epub 2018 Jan 25. PMID 29372461